CLINICAL TRIAL: NCT06278935
Title: Adapting a Lifestyle-based Offloading Intervention in Diabetic Foot Ulcers
Brief Title: Adapting Lifestyle Offloading for DFUs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Tze-Woei Tan, Associate Professor of Clinical Surgery, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APP-24-00887
Record Dates: First submitted 2024-02-16; First posted 2024-02-26 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Foot Ulcer; Diabetic Foot
Keywords: Offloading diabetic foot ulcer; Lifestyle-focused intervention; Occupational therapy; Occupational therapist; Self management
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle-based intervention by an occupational therapist (Experimental): Participants with diabetic foot ulcers will be offered lifestyle-based treatment sessions over telemedicine for up to 8 sessions with a licensed occupational therapist.
  Interventions: Behavioral: Lifestyle-based intervention by an occupational therapist

INTERVENTIONS:
Behavioral: Lifestyle-based intervention by an occupational therapist — Participants with diabetic foot ulcers will be offered lifestyle-based treatment sessions virtually for up to 8 sessions (~8 weeks) with a licensed occupational therapist.

SUMMARY:
The goal of this pilot clinical trial is to develop and test a tailored occupational therapist-led lifestyle-focused intervention to aid patients in improving diabetic foot ulcer care. The main questions it aims to answer are to determine the acceptability and feasibility of taking a tailored lifestyle-focused approach as part of comprehensive diabetic foot ulcer management. Patient participants with DFUs who require offloading treatment will receive the tailored lifestyle-focused self-management intervention.

DETAILED DESCRIPTION:
Diabetic foot ulcers (DFUs) frequently lead to major amputation and mortality. While relieving foot pressure (i.e., offloading) is vital for healing, many patients struggle to adhere to recommended offloading treatments. Participants with DFUs who require offloading treatment will receive the tailored lifestyle-focused self-management intervention. This occupational therapist-led lifestyle-focused intervention will be co-developed with participants, caregivers, family members, and DFU care team members.

Participants with DFUs will be offered lifestyle-based treatment sessions for up to 8 weeks (virtually) with a licensed occupational therapist. Participants will complete pre/post surveys and a subset will take part in an interview to clarify key findings from surveys and obtain patients' perspective of the effectiveness of the intervention. Investigators will also offer focus group interviews to the DFU care team members and occupational therapist to learn their perceptions on the intervention's acceptability, appropriateness, efficiency, and feasibility at the conclusion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Age 21 years or older
* History of active DFU necessitating offloading
* Capacity to provide informed consent
* Access to telehealth (internet connection and equipment)
* Ability to walk independently or with an assistive device
* Self-reported life expectancy of more than one year

Exclusion Criteria:

* Self-reported deafness or blindness
* history of lower extremity amputation besides toes

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction (change from baseline) | Baseline and discharge from OT (3 to 8 weeks)
  Participants will fill out a general satisfaction survey, adapted from and comprising 18 items from a validated measure: Short-Form Patient Satisfaction Questionnaire (PSQ-18). The scale ranges from 1 (strongly agree) to 5 (strongly disagree).

SECONDARY OUTCOMES:
Diabetes distress (change from baseline) | Baseline and discharge from OT (3 to 8 weeks)
  Participants will complete the Type 2 Diabetes Distress Assessment System (T2D-DAS). The T2D-DAS is a validated, multidimensional self-report measure designed to assess diabetes-related distress in adults with type 2 diabetes. It includes 7 domain-specific sources of distress across key areas of diabetes self-management and psychosocial impact (i.e., 7 sources of distress including hypoglycemia, long-term health, health care provider, interpersonal issues, shame or stigma, health care access, and management demands). The T2D-DAS provides a comprehensive profile of diabetes distress. Each item is rated on a 5-point Likert scale ranging from 1 ("Not a problem") to 5 ("A very serious problem"). Subscale scores are calculated as the mean of items within each domain. Higher scores indicate greater diabetes distress.
Offloading knowledge and attitudes (change from baseline) | Baseline and discharge from OT (3 to 8 weeks)
  Participants will complete 41 items of an offloading-specific knowledge and attitudes survey. This survey includes common factors known to influence healing of diabetic foot ulcers (e.g., history of ulcers, access to transportation) and assessment of a person's knowledge of good offloading practices and their attitudes toward those practices. Questions are mixed in style/format, including 5-point Likert (strongly disagree [1] to strongly agree [5]) items such as "My wound does not worry me because it is not painful", yes/no (e.g., "In the past I had a foot wound linked to my diabetes."), and short answer (e.g., "How do you get to the place where you receive treatment for your foot ulcer?"). There is no total score available. Change from baseline in the 27 Likert-scale questions will be assessed individually for each item.
Frequency of DFU-related outcomes | 6-month post-enrollment
  Number of participants with various DFU-related outcomes including DFU healing, minor amputation, major amputation, and ulcer recurrence after healing as extracted from electronic medical record documentation 6 months post-enrollment to the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided